CLINICAL TRIAL: NCT07276958
Title: A Phase 1, Multicenter, Randomized, Placebo-Controlled, Participant-Blind, Single-Ascending Dose Study of LY4298445 in Healthy Participants and an Open-Label Single-Ascending Dose and Multiple-Ascending Dose Study of LY4298445 in Participants With Systemic Lupus Erythematosus or Rheumatoid Arthritis
Brief Title: A Study of LY4298445 in Healthy Participants and Participants With Systemic Lupus Erythematosus (SLE) or Rheumatoid Arthritis (RA)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 27747; J6S-MC-KCAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Systemic Lupus Erythematosus; Rheumatoid Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LY4298445 (Part A1) (Experimental): Single-ascending dose (SAD) of LY4298445 administered subcutaneously (SC) or intravenously (IV) in healthy participants
  Interventions: Drug: LY4298445
- LY4298445 Placebo (Part A1) (Placebo Comparator): SAD of LY4298445 administered SC or IV in healthy participants
  Interventions: Drug: LY4298445
- LY4298445 (Part A2) (Experimental): SAD of LY4298445 administered SC in participants with systemic lupus erythematosus (SLE) or rheumatoid arthritis (RA)
  Interventions: Drug: LY4298445
- LY4298445 (Part B) (Experimental): Multiple-ascending doses (MAD) of LY4298445 administered SC in participants with SLE or RA
  Interventions: Drug: LY4298445
- LY4298445 (Part C) (Experimental): Single dose of LY4298445 administered SC in healthy Japanese and Chinese participants
  Interventions: Drug: LY4298445
- LY4298445 Placebo (Part C) (Placebo Comparator): Single dose of LY4298445 administered SC in healthy Japanese and Chinese participants
  Interventions: Drug: LY4298445

INTERVENTIONS:
Drug: LY4298445 — Administered SC
Drug: LY4298445 — Administered IV
  Arms: LY4298445 (Part A1); LY4298445 Placebo (Part A1)

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of LY4298445 in healthy participants and in participants with systemic lupus erythematosus (SLE) or rheumatoid arthritis (RA). Participation in the study will last up to approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria: Healthy Participants

Healthy participants between the ages of 18 and 55 years.

* Have body weight of at least 50 kilograms (kg) and body mass index (BMI) between 18 and 32 kilogram per square meter (kg/m²), inclusive.

Participants with Systemic Lupus Erythematosus (SLE)

* Are 18 to 75 years of age, inclusive.
* Have body weight between 45 and 145 kg, inclusive, and BMI between 18 and 35 kg/m², inclusive.
* Have a clinical diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria at least 6 months prior to screening.

Participants with Rheumatoid Arthritis (RA)

* Are 18 to 75 years of age, inclusive.
* Have body weight between 45 and 145 kg, inclusive, and BMI between 18 and 35 kg/m², inclusive.
* Have a diagnosis of adult-onset RA for at least 6 months prior to screening, as defined by the 2010 ACR/EULAR classification criteria
* Have Disease Activity Score in 28 joints (DAS28)-high-sensitivity C-reactive protein (hsCRP) greater than or equal to 4.4.
* Have positive test results for rheumatoid factor or anti-citrullinated peptide antibodies
* Have had a history of failure (an inadequate response, intolerance, or loss of response) to at least 2 advanced therapies (biological disease-modifying antirheumatic drug [bDMARD] or targeted synthetic DMARD [tsDMARD]) after failing a conventional synthetic DMARD (csDMARD).

Exclusion Criteria:

* Have known allergies to LY4298445, related compounds, or any components of the formulation
* Are individuals assigned female at birth (AFAB) who are lactating or have a positive pregnancy test at screening or Day -1.
* Have severe active lupus-associated renal disease (lupus nephritis) defined clinically and/or by

  * urine protein/creatinine ratio greater than 200 milligrams per millimole (mg/mmol) (as an estimate of approximate proteinuria greater than 2 reams (g) per day) or
  * an estimated glomerular filtration rate (eGFR) less than 40 milliliters per minute (mL/min)/1.73 m² at screening, as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) 2021.
  * requiring hemodialysis within 6 months prior to screening
* Have active central nervous system lupus as defined by ACR nomenclature for neuropsychiatric lupus syndromes and as captured by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K); seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, and cerebrovascular accident, within 2 months prior to screening
* Have a Class 4 RA according to the ACR revised criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 52
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY4298445 | Baseline up to Approximately Week 57
  PK: AUC of LY4298445
PK: Maximum Concentration (Cmax) of LY4298445 | Baseline up to Week 52
  PK: Cmax of LY4298445
Pharmacodynamic (PD): Degree of Peripheral B Cell Depletion Following Biopsy in Participants | Baseline up to Week 52
  PD: Peripheral B cell depletion

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Nucleus Network, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No